CLINICAL TRIAL: NCT00871923
Title: A Phase II Study to Determine the Efficacy of Tarceva® (Erlotinib Hydrochloride) With Concurrent Whole Brain Radiation Therapy in Patients With Brain Metastases From Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Tarceva With Whole Brain Radiation Therapy - Brain Mets From Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0170; NCI-2012-01649 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Non-small Cell Lung Cancer; Brain Cancer
Keywords: Non-small cell lung cancer; NSCLC; Brain Metastases; Brain Cancer; Lung Cancer; Tarceva; Erlotinib Hydrochloride; OSI-774; Radiation Therapy; Whole Brain Radiation Therapy; WBRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tarceva + RT (Experimental): Tarceva (Erlotinib hydrochloride) + Radiation Therapy. Tarceva 150 mg by mouth every day beginning Day 1. Whole Brain Radiation Therapy (WBRT) for total dose of 3500cGy in 14 daily fractions beginning after Day 6.
  Interventions: Drug: Tarceva (Erlotinib hydrochloride); Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Tarceva (Erlotinib hydrochloride) — 150 mg by mouth every day beginning Day 1.
  Other Names: OSI-774
Radiation: Radiation Therapy — Whole Brain Radiation Therapy (WBRT) for total dose of 3500cGy in 14 daily fractions beginning after Day 6.
  Other Names: RT; XRT; Radiotherapy

SUMMARY:
The goal of this clinical research study is to learn whether Tarceva (erlotinib hydrochloride), when given in addition to whole brain radiation therapy, is better to treat brain metastases in patients with Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
The Study Drugs:

Erlotinib hydrochloride is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take the study drug on Days 1-6 before receiving radiation therapy. You will take 1 pill each day at least 1 hour before or 2 hours after eating. You will take the study drug while you are receiving radiation therapy. You will continue to take the study drug daily after the radiation therapy is complete for as long as the study doctor thinks it is necessary.

You will record at what time each day you take the study drug on a calendar that the will be provided to you. You will bring this calendar with you to each of your study visits.

During the time you are taking the study drug, you must tell the research staff if you have any changes in the drugs that you are taking. If you feel you are having any problems from the study drug before starting radiation therapy, you must tell the study doctor right away.

Radiation Therapy:

After Day 6 of taking the study drug, you will begin radiation therapy. You will receive radiation therapy 1 time each day (Monday through Fridays only) for a total of 14 days.

Once a week during radiation therapy:

* You will have a physical exam.
* You will complete a quality of life questionnaire (at the last week visit)
* You will complete a mini-mental status exam (at the last week visit)
* You will be asked about any changes in the drugs you may be taking
* You will be asked about how you are feeling and any side effects that you may be having
* You will have blood drawn (about 1/2 teaspoon) for lab tests if necessary.

One month after Radiation therapy follow up:

* You will have a follow up visit 1 month after radiation therapy is complete. The study doctor will decide if you will continue to take the study drug at the follow-up visit. The following tests and procedures will be performed:
* You will have a physical exam.
* You will have an MRI or CT of the brain.
* Your vital signs will be recorded.
* You will complete a quality of life questionnaire.
* You will complete a mini-mental status exam.
* You will be asked about any changes in the drugs you may be taking.
* You will be asked about how you are feeling and any side effects that you may be having.
* You will have blood drawn (about 1/2 teaspoon) for lab tests if necessary.

Follow-up Visits (While on Tarceva):

If, at the end-of-study visit, the doctor decides that you will continue to take the study drug, you will have a follow-up visit with the research nurse 1 time each month. At these visits, the following tests and procedures will be performed:

(If unable to return to MDACC, this visit will be conducted over the telephone and arrangements will be made to mail study Tarceva medication.)

* Your medical history will be reviewed.
* You will receive a 30-day supply of the study drug.
* You will bring in your study drug calendar for the nurse to review.
* You will be asked about how you are feeling and any side effects that you may be having.
* You will also be asked about any changes in the drugs you may be taking.
* Blood (about 1/2 teaspoon) may be drawn for routine tests.

The following tests and procedures will be performed every 3 months:

* You will have a physical exam.
* You will have an MRI or CT of the brain
* Your vital signs will be recorded.

Follow up visit (Discontinuation of Study Drug):

You will have a follow up visit with the research nurse 1 month after your last dose of the study drug, and the following will be performed:

(If unable to return to MDACC, this visit will be conducted over the telephone and arrangements will be made to have the study Tarceva medication and medication diary returned by mail.)

* Your medical history will be reviewed.
* You will be asked about how you are feeling and any side effects that you may be having.
* You will return your study drug calendar and any remaining Tarceva tablets to the research nurse.
* You will also be asked about any changes in the drug you may be taking
* Your vital signs will be recorded.

The following tests and procedures will be performed every 3 months (off Tarceva) for the first 2 years then every 6 months thereafter:

* You will have a physical exam.
* Your medical history will be reviewed.
* You will have an MRI or CT of the brain
* If you are unable to return for your follow up visits due to physical conditions, you will be contacted by phone.

Duration of Study Treatment:

You will remain on study for as long as the study doctor thinks you are benefitting from the study drug. You will be taken off study treatment early if the disease gets worse, you experience intolerable side effects, or your doctor thinks that it is no longer in your best interest to continue to receive treatment on this study.

This is an investigational study. Erlotinib hydrochloride is FDA approved and commercially available. It has not been FDA approved to treat NSCLC that has spread to the brain.

Up to 20 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of non-small cell lung cancer
2. Patients who have been treated in the past with stereotactic radiosurgery, stereotactic radiotherapy, GliaSite or surgical resection will be allowed to enroll in this study
3. A diagnostic contrast-enhanced MRI or CT scan must be performed, demonstrating brain metastases
4. Age 18-70
5. Patients must have KPS >/= 70
6. Patients cannot be treated on any other treatment related protocols within 30 days prior to study entry or during participation in the study
7. No uncontrolled or symptomatic major medical illnesses or psychiatric impairments, such as Alzheimer's or schizophrenia
8. Screening Clinical Laboratory Values: ANC >1500/ul, Platelets >80,000/ul, baseline AST and/or ALT within normal limits (within 30 days of starting protocol treatment)
9. All women of childbearing potential (A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]) and male participants must practice effective contraception (abstinence, oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study.
10. Continued from #10: All women of child-bearing potential must have a negative serum pregnancy test and practice birth control while on study.
11. Patients must provide verbal and written informed consent to participate in the study.

Exclusion Criteria:

1. Prior cranial radiation therapy, other than stereotactic radiosurgery, Stereotactic Radiotherapy or GliaSite.
2. Patients with known Acquired Immune Deficiency (AIDS), as regimens with tyrosine kinase inhibitors may pose a safety risk related to excess toxicity or interference with anti-viral effectiveness
3. Women who are pregnant or lactating, due to possible adverse effects on the developing fetus or infant due to study drug
4. Patients with active connective tissue disorders, such as lupus or scleroderma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-03-26 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Welsh, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Welsh JW, Komaki R, Amini A, Munsell MF, Unger W, Allen PK, Chang JY, Wefel JS, McGovern SL, Garland LL, Chen SS, Holt J, Liao Z, Brown P, Sulman E, Heymach JV, Kim ES, Stea B. Phase II trial of erlotinib plus concurrent whole-brain radiation therapy for patients with brain metastases from non-small-cell lung cancer. J Clin Oncol. 2013 Mar 1;31(7):895-902. doi: 10.1200/JCO.2011.40.1174. Epub 2013 Jan 22. PMID 23341526
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 44 patients were consented to this study, but 1 patients withdrew consent prior to protocol treatment. 43 patients was treated under this protocol.
Groups:
- Phase II Tarceva for Brain Metastases in NSCLC: Patients were treated with Tarceva 150mg PO daily. On day 7, whole brain radiation 3000cGy/10. remained on Tarceva until disease progression/toxicity
Period: Overall Study
Arm/Group | Phase II Tarceva for Brain Metastases in NSCLC
Started | 44
Completed | 42
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 43 out of 44 patients was were consented and treated under this protocol. 1 patients withdrew consent prior to protocol treatment.
Arm/Group | Phase II Tarceva for Brain Metastases in NSCLC
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 59 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 32
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 42
  Mexico | 1
Karnofsky Performance Score (KPS) [Count of Participants; unit: Participants] — The KPS ranking runs from 100 to 0, where 80: Normal activity with effort; some signs or symptoms of disease. 70: Cares for self; unable to carry on normal activity or to do active work. The KPS was to allow physicians to evaluate a patient's survival. The higher KPS scores, the better treatment outcome.
  Participants
    KPS≥ 80 | 29
    KPS≤ 70 | 14
Tumor Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 32
  Other | 9
  Squamous | 2
Smoking History [Count of Participants; unit: Participants]
  Never | 11
  Prior | 26
  Current | 5
  Unknown | 1
Previous Therapy [Count of Participants; unit: Participants]
  Yes | 29
  No | 14
Number of Brain Metastases [Count of Participants; unit: Participants]
  0-3 | 19
  4 -10 | 16
  >10 | 8

OUTCOME MEASURES:

1. Primary Outcome: Median Survival
Description: Median Survival will be estimated using the method of Kaplan and Meier (1958) using the intent-to-treat principle.
Time Frame: End-of-study visit 1 month after radiation therapy completed, and follow-up visits every 3 months, assessed up to 2 years.
Population: Twenty patients from University of Arizona and 20 patients at MDACC for a total of 40 patients were combined for statistical analysis for Median Survival. We excluded 4 MDACC patients because: 1 patients withdrew consent prior to protocol treatment, I patient death during radiotherapy, 2 patients early death without follow-up data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II Tarceva for Brain Metastases in NSCLC
Number analyzed (Participants) | 40
months | 11.8 [7.4 to 19.1]

2. Secondary Outcome: Number of Participants With Overall Survival
Description: Overall Survival will be estimated using the method of Kaplan and Meier (1958) using the intent-to-treat principle. The participants overall survival measured at 6 month, 1-year and 2 years.
Time Frame: From date of registration until the date of first documented death or lost to follow up, whichever came first, assessed up to 2 years.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Tarceva for Brain Metastases in NSCLC
Number analyzed (Participants) | 40
Participants
  6-month | 27
  1-year | 20
  2-year | 7

ADVERSE EVENTS:
Time Frame: From date of protocol registration until the date of documented development of adverse events (AEs) , assessed up to 2 years.
Arm/Group | Phase II Tarceva for Brain Metastases in NSCLC
All-Cause Mortality (participants affected / at risk) | 36/43
Serious Adverse Events (participants affected / at risk) | 26/43
Other Adverse Events (participants affected / at risk) | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II Tarceva for Brain Metastases in NSCLC (N=43)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1)
Acne Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Dehydration (Gastrointestinal disorders) | 6 (7)
Fatigue (Congenital, familial and genetic disorders) | 6 (7)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Upper GI Bleed (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Increased AST/ALT (Hepatobiliary disorders) | 2 (2)
Increased bilirubin (Hepatobiliary disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Anorexia (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspepsia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspenea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Weight Loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT00871923/Prot_SAP_000.pdf